CLINICAL TRIAL: NCT01643551
Title: Neuron Specific Enolase in Ventricular Assist Device Recipients
Acronym: NSE-LVAD
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1204M12861
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Advanced Heart Failure; Left Ventrucular Assist Device
Keywords: Heart Failure; Left Ventricular Assist Device; Reperfusion Injury; Neuron Specific Enolase
MeSH Terms: conditions — Heart Failure; Reperfusion Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LVAD Group: 18 years and older Planning to undergo VAD implantation
- Cardiac Surgery Group: 18 years or older Planning to undergo valve or coronary bypass surgery

SUMMARY:
An observational study of neuron specific enolase, as a marker of reperfusion injury, in LVAD recipients before and following VAD implantation.

DETAILED DESCRIPTION:
Patients eligible for left ventricular assist device (LVAD) typically have severe heart failure, which is characterized by poor cardiac output. The relatively abrupt increase in cardiac output that follows implant of a LVAD may cause reperfusion injury. Furthermore, selected patients may have particularly severe consequences of such injury, including refractory acidosis and vasoplegia. Neuron specific enolase (NSE) has been established as a biomarker of reperfusion injury. We hypothesize that changes in NSE following LVAD will be greater than the changes in NSE noted in a control population of patients undergoing non-VAD cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

Group 1 - Pre-VAD implantation patients

* 18 years and older
* lanning to undergo VAD implantation Group 2 Cardiac Surgery Comparison Group
* 18 years or older
* Planning to undergo valve or coronary bypass surgery

Exclusion Criteria:

* Acute cerebrovascular infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiovascular Surgical candidates from outpatient cardiology clinic or inpatient service.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Neuron-Specific Enolase | Pre and post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Eckman, MD, Principal Investigator — University of Minnesota; Demitri Yannopoulos, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota, United States